CLINICAL TRIAL: NCT05985798
Title: Sintilimab, Bevacizumab Plus TACE Versus Lenvatinib Plus TACE for Advanced Stage Hepatocellular Carcinoma: A Randomized Controlled Trial
Brief Title: Sintilimab+Bevacizumab+TACE vs. Lenvatinib+TACE for Advanced HCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Affiliated Hospital of Guangdong Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Lecong Hospital, Shunde District, Foshan (Unknown); First People's Hospital of Foshan (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-13
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sin-Bev-TACE (Experimental): Sintilimab, bevacizumab plus TACE
  Interventions: Drug: Sin-Bev-TACE
- Len-TACE (Active Comparator): Lenvatinib plus TACE
  Interventions: Drug: Len-TACE

INTERVENTIONS:
Drug: Sin-Bev-TACE — Sintilimab (200mg I.V. q3w) and bevacizumab (7.5mg/kg I.V. q3w) are administered at 3-7 days after the first TACE. The study treatment of sintilimab and bevacizumab will last up to 24 months. TACE can be repeated on demand.
  Arms: Sin-Bev-TACE
Drug: Len-TACE — Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd will be started at 3-7 days after the first TACE. TACE will be repeated on demand.
  Arms: Len-TACE

SUMMARY:
This study is conducted to evaluate the efficacy and safety of sintilimab, bevacizumab plus TACE (Sin-Bev-TACE) compared with lenvatinib plus TACE (Len-TACE) for patients with advanced stage hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a multicenter, prospective and randomized controlled trial to evaluate the efficacy and safety of Sin-Bev-TACE versus Len-TACE for patient with advanced HCC.

258 patients with advanced HCC (BCLC C stage) will be enrolled in this study. The patients will receive either sintilimab and bevacizumab (Sin-Bev) or lenvatinib (Len) after first TACE using an 1:1 randomization scheme. In the Sin-Bev-TACE arm, sintilimab (200mg I.V. q3w) and bevacizumab (7.5mg/kg I.V. q3w) will be started at 3-7 days after the first TACE. In the the Len-TACE arm, lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd will be started at 3-7 days after the first TACE.

TACE will be repeated on demand based on the evaluation of follow-up laboratory and imaging examination. Sintilimab and bevacizumab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Lenvatinib will last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. In the Sin-Bev-TACE arm, patients will be allowed to have sintilimab or bevacizumab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

The primary end point of this study is overall survival (OS). The secondary endpoints are progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Advanced HCC (BCLC stage C) with diagnosis confirmed pathologically or clinically
* Disease amenable to TACE
* No prior systemic therapy, TACE, transcatheter arterial radioembolization (TARE), transcatheter arterial embolization (TAE), hepatic arterial infusion chemotherapy (HAIC) or radiation therapy for HCC
* Child-Pugh class A
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Life expectancy of at least 3 months
* At least one measurable intrahepatic lesion
* Adequate organ and hematologic function
* Patients with active hepatitis B are allowed, but they need to receive antiviral treatment to achieve a HBV DNA<10^2 IU/mL
* Patients with hepatitis C need to finish the anti-HCV treatment

Exclusion Criteria:

* Tumor thrombus involving main portal vein or both the first left and right branch of portal vein
* Vena cava invasion
* Central nervous system metastasis
* History of hepatic encephalopathy
* History of organ and cell transplantation
* Uncontrolled ascites, hydrothorax or pericardial effusion
* Prior esophageal and/or gastric varices bleeding within 6 months prior to initiation of study treatment
* Presence of known severe (G3) varicose veins in endoscopy within 3 months before the first dose. Evidence of portal hypertension (including the finding of splenomegaly in imaging studies) with a high risk of bleeding assessed by the investigator
* Presence of any life-threatening bleeding events within the past 3 months, including the need for transfusion, surgery or local treatment, and continuous medication therapy
* Any arterial or venous thromboembolic events within 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient cerebral ischemic attack, pulmonary embolism, deep vein thrombosis, or any other history of serious thromboembolism. Presence of implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis, barring stable thrombosis following the conventional anticoagulation treatment. Prophylactic use of low-dose low-molecular-weight heparin (e.g., enoxaparin 40 mg/day) is permitted.
* A 10-day consecutive dosing of aspirin (> 325 mg/day) or other drugs, e.g., dipyridamole and clopidogrel, known to inhibit the platelet function within 2 weeks before the first dose
* Uncontrolled hypertension after the optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
* Symptomatic congestive cardiac failure (NYHA Class II-IV). Symptomatic or poorly controlled arrhythmia. History of congenital long QT syndrome or corrected QTc > 500 ms (calculated using Fridericia formula) during screening
* Serious hemorrhagic tendency or coagulopathy, or currently receiving thrombolytic therapy
* History of gastrointestinal perforation and/or fistula, history of bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection accompanied with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within the past 6 months
* History or current experience of pulmonary fibrosis and such lung diseases as interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severely impaired lung function
* Active tuberculosis (TB), currently receiving anti-tuberculosis treatment or received such treatment within 1 year before the first dose
* Human immunodeficiency virus (HIV) infected (HIV 1/2 antibody positive) and known syphilis infection requiring treatment
* Active or poorly clinically controlled serious infections. Severe infections within 4 weeks before the first dose, including but not limited to hospitalization caused by infection, bacteremia, or severe pneumonia complication
* Presence of active autoimmune diseases requiring systemic treatment (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first dose. Use of alternative therapies (e.g., thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is permitted. Known history of primary immunodeficiency diseases. For patients with positive autoimmune antibodies only, they should be assessed by the investigator to determine whether they had an autoimmune disease
* Receipt of immunosuppressants within 4 weeks before the first dose, excluding local glucocorticoids administered by nasal, inhaled, or other topical routes, or systemic glucocorticoids of physiological doses (no more than 10 mg/day of prednisone or equivalents), while the temporary use of glucocorticoids for preventing allergies or treating dyspneic symptoms of such diseases as asthma and chronic obstructive pulmonary disease is permitted
* Receipt of major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose or having unhealed wounds, ulcers, or fractures. Receipt of tissue biopsy or other minor surgeries within 7 days before the first dose, barring venipuncture and catheterization for intravenous infusion.
* Receipt of systemic treatment with traditional Chinese medicines with cancer indications or immunomodulators (including thymosin, interferon, and interleukin, barring local use for controlling pleural fluid or ascites) within 2 weeks before the first dose
* History of malignancy other than HCC
* Known hypersensitivity to any ingredients in sintilimab, bevacizumab and lenvatinib preparations or previous severe hypersensitivity reactions to other monoclonal antibodies
* Pregnant or breastfeeding female patients
* Acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may lead to the following consequences: increased study participation or drug-related risks, or interference with interpreting trial results, and considered ineligible for participating in the trial by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 4 years
  The time from date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 4 years
  The time from date of randomization until the first occurrence of disease progression or death due to any cause, whichever occurs first.
Objective response rate (ORR) | 4 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR).
Disease control rate (DCR) | 4 years
  The proportion of patients with the best response of CR, PR, or stable disease (SD).
Adverse Events (AEs) | 4 years
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China